CLINICAL TRIAL: NCT01426620
Title: Salvage Therapy With Docetaxel and Blueberry Powder in Non-Small Cell Lung Cancer
Brief Title: Standard Chemotherapy With Blueberry Powder in Non-Small Cell Lung Cancer
Acronym: BIT-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Goetz Kloecker, Associate Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC-LUN-BIT-2
Record Dates: First submitted 2011-08-27; First posted 2011-08-31 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; blueberry; salvage therapy; docetaxel; non-small cell lung cancer; second-line; polyphenol
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blueberry powder (Experimental): This is a two-part open-label clinical trial of blueberry powder administered to patients with stage IV NSCLC in combination with docetaxel as a second line treatment. Patients will initially be enrolled in part 1 of the study, which is the feasibility/toxicity evaluation section of the study. Once the part I enrollment is completed, the patients will be enrolled in part 2 of the study.
  Interventions: Dietary Supplement: Blueberry powder

INTERVENTIONS:
Dietary Supplement: Blueberry powder — The intervention consists of 2-3 packages (15 grams per package) of lyophilized blueberry powder, taken daily after mixing with natural yogurt, milk, water, or juice in combination with set dosage of docetaxel (35 milligrams per meter squared) administered intravenously every week for 4 cycles, 21-day cycles.

SUMMARY:
This phase II trial will evaluate phyto-therapy's, in the form of blueberry powder, synergistic effect on second-line therapy for non-small cell lung cancer (NSCLC). The proposition is that the addition of blueberry polyphenolics to routine docetaxel therapy will have a significant, positive effect in the response rate and overall survival.

DETAILED DESCRIPTION:
This study is designed to evaluate the feasibility of using blueberry powder (rich in anthocyanidins) as an adjunct therapy with the conventional chemotherapy drug paclitaxel/docetaxel for treatment of NSCLC. The study is based on information from published studies in which blueberry anthocyanidins (bioflavonoids which give blueberries their color) have been shown to regulate a vast array of molecular targets, and on our own exciting and compelling preliminary data showing that blueberry anthocyanidins elicited potent synergistic chemo-sensitizing effects in two highly aggressive non-small cell lung cancer (NSCLC) cell lines.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to screening
2. Male or female patients, age ≥ 18 years
3. Histologically or cytologically confirmed diagnosis of NSCLC
4. Stage IV disease (including patients with pleural effusion previously classified as Stage IIIB)
5. All of the following if patient has had prior radiation therapy:

   * lesion(s) used for determination of response were not previously irradiated or have increased in size since the completion of radiotherapy
   * the patient has recovered from any acute effects of the radiotherapy
   * radiotherapy was completed at least 4 weeks prior to screening
6. Part 1: Have at least non-measurable evaluable disease (e.g., lesions which are smaller than the minimum size required for measurability; other non-measurable lesions such as bone metastases, malignant pleural effusion)
7. Part 2: Have measurable disease, defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded) as > 10 millimeters (mm) on cross-sectional imaging (where the CT slice thickness is no greater than 5 mm) or at least 20 mm by standard techniques; positron emissions tomography [PET] and ultrasound are not permitted methods for tumor measurements under this protocol.
8. Performance status of 0 or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale
9. Have an estimated life expectancy of at least 12 weeks
10. Adequate organ function within 14 days prior to first berry powder dose or docetaxel whichever occurs first, including the following - absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, hemoglobin ≥ 9 g/dL (≥ 5.6 mmol/L), patients may receive packed red blood cells (RBC) transfusion to achieve this level at the discretion of the investigator, total bilirubin < 1.5 x upper limit of normal (ULN) unless elevated secondary to conditions such as Gilbert's Disease, aspartate aminotransferase (AST) < 3 x ULN (< 5 x ULN in the presence of hepatic metastases), alanine aminotransferase (ALT) < 3 x ULN (< 5 x ULN in the presence of hepatic metastases), alkaline phosphatase < 3.0 x ULN, calculated creatinine clearance ≥ 60 mL/min per Cockcroft and Gault formula
11. Satisfy one of the following:

    * Females: non-pregnant and non-lactating; surgically sterile, post-menopausal, or patient/partner compliant with a reliable contraceptive regimen, as determined by the Investigator, for 4 weeks prior to screening. Patients of reproductive potential must test negative for pregnancy at screening and must agree to use a reliable method of birth control during the study period
    * Males: surgically sterile or patient/partner must agree to use a reliable contraceptive method, as determined by the Investigator, during the study period
    * The patient is willing and able to comply with the study visit schedule and procedures, and has geographical proximity (Investigator's discretion) that allows follow-up specified by the protocol
    * For Part 1: have discontinued all prior chemotherapies, biological therapies, and other investigational therapies for cancer for at least 4 weeks (6 weeks for mitomycin-C or nitrosoureas) prior to study treatment and have recovered from the acute effects of therapy

Exclusion Criteria:

1. Part 1: More than one prior chemotherapy (single biological therapy, i.e., Erlotinib not included) regimens (approved or experimental) for NSCLC, not counting adjuvant and neoadjuvant treatment. A regimen is defined as two or more consecutive cycles of treatment. Part 2: Any prior chemotherapy or biological therapy (approved or experimental) for NSCLC including adjuvant and neoadjuvant treatments
2. Treatment with another investigational drug, biological agent, or device within 4 weeks (6 weeks for biological agents) before screening or 5 half-lives of study agent, whichever is longer
3. Patients with treated or untreated parenchymal brain metastases or leptomeningeal disease. Brain imaging is required for symptomatic patients to rule out brain metastases, but is not required in asymptomatic patients
4. Patients with known pericardial effusion
5. Patients with active infection or serious concomitant systemic disorder (for example, heart failure) incompatible with the study (at the discretion of the Investigator)
6. Presence or history of malignancy other than NSCLC, carcinoma in situ of the cervix, or non-melanoma skin cancer. In the case of other malignancies, patients may be considered for participation if the prior malignancies were diagnosed and definitively treated at least two years previously with no subsequent evidence of recurrence.
7. Presence of an underlying disease state associated with active bleeding
8. Concurrent treatment with other anticancer drugs
9. Pre-existing peripheral neuropathy ≥ Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE) Grade 2
10. Planned concomitant participation in another clinical trial of an experimental agent, vaccine, or device
11. Patients with any other medical conditions that in the opinion of the Investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in or completing the study
12. Allergy to berries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients successfully completing the entire treatment plan | 2 years after study enrollment
  Completion of treatment plan by 10 patients. Feasibility and toxicity for the study will be evaluated in Part 1 of the study based on 10 patients completing the treatment plan (20 if 2 of the initial 10 patients develop toxicities).
Clinical Response Rate | 16 months after last treatment
  Clinical response (complete, partial and sustained) rates will be evaluated using Response Evaluation Criteria in Solid Tumor (RECIST) Guidelines (version 1.1)

SECONDARY OUTCOMES:
Cumulative number of grade 3 or 4 toxic events | 2 years after study enrollment
  The cumulative number of toxic grade 3 or 4 events after each person is treated will be compared to the boundary outlined in the protocol. If the cumulative number of toxic events produces enough evidence to conclude that the true toxicity rate is greater then or equal to 33% (Pt0 = 0.33), then the trial will be stopped early for safety reasons.
Progression-free survival (PFS) time | 16 months after last treatment
  Progression-free survival time defined as the time from enrollment until the first indication of disease progression or death due to any cause. Progression will be determined based on radiological measurements using RECIST criteria.
Overall Survival (OS) | 2 years after time of enrollment of last participant
  Overall Survival (OS) - time will be determined as the time from enrollment until death or last follow-up evaluation.
Change in biomarker levels, measured by blood tests taken throughout the study | 2 years after study enrollment
  The changes in biomarker levels and their association with response assessments will be studied.
Quality of Life FACT-L measurement | 2 years after study enrollment
  Functional Assessment of Cancer Therapy-Lung(FACT-L) questionnaire will be used to evaluate and measure quality of life.
Measure the change in berry polyphenolic levels by blood tests throughout the study | 2 years after study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Goetz H Kloecker, MD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States